CLINICAL TRIAL: NCT03992586
Title: Effect of Rose-colored Glass on Mood: A Randomized Clinical Trial
Brief Title: Effect of Rose-colored Glass on Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Center for Dermatology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RCG101
Record Dates: First submitted 2018-08-14; First posted 2019-06-20 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Mood

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pink lenses (Experimental): Pink-colored lenses
  Interventions: Other: Wearing pink glasses
- Clear lenses (Placebo Comparator): Clear lenses
  Interventions: Other: Wearing clear glasses

INTERVENTIONS:
Other: Wearing pink glasses — Wearing pink-colored lenses
  Arms: Pink lenses
Other: Wearing clear glasses — Wearing clear glasses
  Arms: Clear lenses

SUMMARY:
Decades of psychological research has highlighted the impact of visual perception on mood and happiness. The investigators hypothesized that literally seeing the world through rose colored glasses may have an effect on perception, mood, and happiness. After cataract surgery, which classically increases the vividness of perceived colors, patients report significant satisfaction. The investigators therefore sought to explore whether using pink colored lenses leads to a measurable impact on outcomes.

DETAILED DESCRIPTION:
A randomized controlled clinical trial design will be performed. Subjects will be randomized for either pink lenses (treatment group) or clear lenses (placebo group).

Subjects will be asked to wear the assigned glasses throughout the day during the course of the trial. Glasses will not be work while driving at night.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years of age.

Exclusion Criteria:

* Subjects who wear glasses on a regular basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Anxiety Scores on the Visual Analogue Scale at 1 week | 1 week
  Scale range 0-100, higher values represent more anxiety

SECONDARY OUTCOMES:
Change from baseline in Mood Scores on the Visual Analogue Scale | 1 week
  Scale range 0-100, higher values represent more sadness
Change from baseline in Happiness Scores on the Visual Analogue Scale | 1 week
  Scale range 0-100, higher values represent more happiness
Change from baseline in the Center for Epidemiological Studies Depression Scale score | 1 week
  Scale range 0-60, higher values suggest more depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kantor, MD, Principal Investigator — Florida Center for Dermatology
Locations (1):
- St Vincent's Medical Center, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data are available to other researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data are available to other researchers upon reasonable request.
Access Criteria: Data are available to other researchers upon reasonable request.